CS

Da: clara santavenere clarasantavenere@gmail.com
Oggetto: Re: Richiesta parere di competenza da parte del CE

Data: 8 giugno 2022, 09:20

A: Claudio Celentano celentanoclaudio70@gmail.com

Cc: Segreteria Amministrativa Comitato Etico comitatodietica@unich.it

Gent.mo.

la presente per comunicarle che la pratica in questione è di non competenza del CE che, pertanto, non esprimerà parere a riguardo.

Restando a disposizione, porgo cordiali saluti dott.ssa Clara Santavenere Segreteria tecnico-amministrativa Comitato Etico provv. Ch-Pe

Il giorno mar 7 giu 2022 alle ore 21:15 Claudio Celentano <<u>celentanoclaudio70@gmail.com</u>> ha scritto: Alla C.A. Comitato di Etica

Si allega protocollo di studio legato alla didattica su medici specialisti e specializzandi nella gestione delle emergenze ostetriche su manichini ad alta e bassa fedeltà, al fine di conoscere se tale protocollo necessita di parere da parte del CE a fini di ricerca.

Con osservanza

Claudio Celentano, MD